CLINICAL TRIAL: NCT00778947
Title: Comparison of Harmonic Scalpel to Conventional Diathermy in Free Tissue Transfer for Breast Reconstruction
Brief Title: Single Centre Study to Compare Harmonic Scalpel to Conventional Diathermy in Free Tissue Transfer Breast Reconstruction
Acronym: HARMONIC001
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study abandoned and was never started
Sponsor: St Andrew's Centre for Plastic Surgery (Other)
Responsible Party: Mr V Ramakrishnan, Consultant Plastic Surgeon, St. Andrew's Centre for Plastic Surgery, Broomfield Hospital, Chelmsford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Harmonic Scalpel HARMONIC 001
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2008-10

CONDITIONS: Breast Reconstruction
Keywords: Breast Reconstruction; Halmonic Scalpel; diathermy; Free Tissue Transfer
MeSH Terms: conditions — Fever | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Harmonic Synergy Dissecting Hook (Harmonic Scalpel)
- 2 (Active Comparator)
  Interventions: Procedure: Electrocautery Diathermy

INTERVENTIONS:
Procedure: Harmonic Synergy Dissecting Hook (Harmonic Scalpel) — Harmonic Synergy Dissecting Hook (Harmonic Scalpel) uses ultrasound waves to coagulate and cut in surgery. It is available on the market, holds a CE mark and is coded as a Class IIb medical device.
  Arms: 1
Procedure: Electrocautery Diathermy — Electrosurgery uses high temperatures (150-400oC) and causes obliterative coagulation. Diathermy is the use of high frequency electric current to produce heat. In surgery it is used to cut or destroy tissue and/or to produce coagulation. The electrical frequency produced in diathermy is in the range of 300kHz to 3MHz.
  Arms: 2

SUMMARY:
The purpose of this single centre study is to evaluate whether the use of Harmonic Synergy Dissecting Hook (Harmonic Scalpel) in breast reconstruction surgery is superior to conventional diathermy in terms of improving ease and speed of perforator dissection, reducing postoperative pain, days of hospital stay and time taken to return to daily activities.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 18 and 80 years old
2. Able to comprehend, follow, and provide written informed consent.
3. Willingness to comply with study requirements including follow-up visits

Exclusion Criteria:

1. Patients who have a pacemaker
2. Pregnant or breast feeding females.
3. General contraindication for surgery as deemed by the PI (e.g. physically unfit)
4. Patients who smoke
5. Diabetic patients
6. Patients who are receiving permanent analgesics
7. Patients receiving anti-coagulation therapy.
8. Patients with a physical or psychological condition which would impair participation in the study.
9. Participation in any other device or drug study within 90 days prior to enrollment.
10. Planned participation in any other medical device study during the timeframe of this study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
The speed of flap harvest measured as the time from "knife to skin" to the flap being removed from the patient. | At surgery

SECONDARY OUTCOMES:
Ease of flap harvest: the subjective opinion of the surgeon based on structured questionnaire | At surgery
Post operative pain, based on the visual analogue scale at 3, 6, 12 and 24 weeks post operatively. | 3, 6, 12 and 24 weeks post operation
Rates of post operative infection | post operation for 6 months
Incidence of abdominal (donor site) wound dehiscence | post operation for 6 months
Bleeding complications | intra operation and for 6 months post op
Return to theatre | post operation for 6 months
Incidence of seroma | post operation for 6 months
Post operative drainage from the wound | post operation for 6 months
Impact on daily activities (SF-36 Questionnaire) at 3, 6, 12 and 24 weeks post operatively | 3, 6, 12, and 24 weeks post operation
Number of days of hospitalisation | post operation for 6 months
Re-operation required | post operation for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: V Ramakrishnan, Principal Investigator — St Andrew's Centre for Plastic Surgery
Locations (1):
- St. Andrew's Centre for Plastic Surgery, Broomfield Hospital,, Chelmsford, United Kingdom